CLINICAL TRIAL: NCT05500053
Title: A Study of the Characteristics of Patients Diagnosed With Recurrent Symptomatic Genital Herpetic Disease
Status: Completed | Type: Observational
Sponsor: Rational Vaccines Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: RVx-001-PSS
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Genital Herpes; Patient Engagement
MeSH Terms: conditions — Herpes Genitalis; Patient Participation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determine the baseline characteristics of patients who have recurrent symptomatic genital herpetic disease Determine the acceptance to patients of clinical trial procedures Determine interest in participation in genital herpes vaccine trials

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign the informed consent document.
* Patient confirmation of a diagnosis of HSV-2 infection at least 2 years prior to inclusion. Laboratory confirmation is not required.
* Symptomatic recurrent genital herpetic disease for >2 years supported by compatible clinical history

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria for the study
* Subjects who are unable to provide legally effective informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with recurrent symptomatic of genital herpes
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Baseline characteristics of patients who have recurrent symptomatic genital herpetic disease | day of questionnaire
  To determine using a questionnaire
  * number of annual outbreaks of patients who have recurrent symptomatic genital herpetic disease
  * number of patients using suppressiv antiviral therapy
  * number of patients using antivirals for the treatment of outbreaks
  * number of patients using symptomatic therapy other than antivirals
Acceptance to patients of clinical trial procedures | day of questionnaire
  To determine using a questionnaire
  - the acceptance to patients of clinical trial procedures
Interest in participation in genital herpes vaccine trials | day of questionnaire
  To determine using a questionnaire the number of patients interested in participation in genital herpes vaccine trials

CONTACTS AND LOCATIONS:
Overall Officials: Rajul Patel, Principal Investigator — Solent NHS Trust
Locations (1):
- Solent NHS Trust, Southampton, UK, United Kingdom